CLINICAL TRIAL: NCT00770874
Title: Phase III Study of S-1 + Cisplatin Compared With Single-agent Cisplatin in Stage IVB, Recurrent, or Persistent Carcinoma of the Cervix
Brief Title: Phase III Study of S-1 + Cisplatin vs Cisplatin in Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10020380
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — S 1 (combination); Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): S-1 + Cisplatin (arm A)
  Interventions: Drug: S-1 + Cisplatin (arm A)
- 2 (Active Comparator): Cisplatin (arm B)
  Interventions: Drug: Cisplatin (arm B)

INTERVENTIONS:
Drug: S-1 + Cisplatin (arm A) — S-1 will be administered orally, twice daily from Day 1 through Day 14 followed by a recovery period from Days 15 through Day 21. Initial dose of S-1 will be determined according to the patient's body surface area (80 to 120 mg/day). On Day 1, Cisplatin 50 mg/m2 will be administered intravenously (IV). This regimen is to be repeated every 3 weeks.
  Arms: 1
Drug: Cisplatin (arm B) — Cisplatin 50 mg/m2 will be administered intravenously (IV) on Day 1, repeated every 3 weeks.
  Arms: 2

SUMMARY:
This study is an open-label, multicenter, multinational, two-arm, parallel randomized Phase 3 study evaluating the efficacy and safety of S-1+Cisplatin versus single-agent Cisplatin in patients with stage IVB, recurrent or persistent carcinoma of the cervix.

DETAILED DESCRIPTION:
Japanese phase II study of S-1 in cervical cancer suggested promising response rate and good tolerability. Since recommended chemotherapy for metastatic or recurrent cervical carcinoma is either single-agent Cisplatin or Cisplatin-based combination chemotherapy, this is designed to evaluate the efficacy and safety of S-1 in combination with Cisplatin compared with single-agent Cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven cervical carcinoma (All histological subtype will be included).
* Patients who have stage IVB, recurrent or persistent disease.
* Patients who are not amenable to curative treatment with surgery and/or radiotherapy.
* Patients who have not received chemotherapy or chemoradiotherapy after diagnosis of recurrent, persistent, or stage IVB disease.
* If the patient have received chemotherapy, radiotherapy or chemoradiotherapy as previous treatment, following interval must have elapsed from the last administration of treatment:

  1. Chemotherapy: 21 days
  2. Radiotherapy: 21 days*
  3. Chemoradiotherapy: 42 days*

If there have been residual disease in previously irradiated field and without disease progression since the (chemo) radiotherapy, 90 days must have elapsed after the last administration of irradiation.

* Patients who have adequate hematologic, hepatic and renal functions as defined below:

  * Hemoglobin: ≥ 8.0 g/dL
  * Neutrophil count: ≥ 2,000/mm^3
  * Platelet count: ≥ 100,000/mm^3
  * Total serum bilirubin: ≤ 1.5 times the upper limits of normal (ULN)
  * AST (GOT), ALT (GPT): ≤ 2.5 times the ULN. If abnormal values are associated with hepatic metastasis: ≤ 5.0 times the ULN
  * Serum creatinine: ≤ ULN or creatinine clearance: ≥ 50 ml/min
* Patients who have an ECOG performance status : 0-1.
* Age: ≥ 20 years old.
* Patients who can take pills orally.
* Patients who signed the written consent form.

Exclusion Criteria:

* Patients who have known hypersensitivity to 5-FU or Cisplatin.
* Patients who are receiving concomitant treatment with drugs interacting with S-1.
* Patients who are receiving concomitant treatment with drugs interacting with Cisplatin.
* Patients who were administered other investigational products within 30 days before the initiation of study treatment.
* Patients who were previously treated with S-1.
* Patients who had received platinum-containing chemotherapy or chemoradiotherapy and whose disease progressed during the therapy.
* Patients who suffer from active infection (e.g. fever ≥ 38°C).
* Patients who have serious complications.
* Patients with bleeding which requires hemostasis treatment.
* Patients with bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage.
* Patients with uncontrolled pleural effusion and/or ascites requiring drainage at least twice a week.
* Patients with symptomatic brain metastasis or history of brain metastasis.
* Patients who have unmanageable bowel movement (ex. Watery stool, chronic constipation).
* Patients with active double cancer.
* Patients who are pregnant or lactating.
* Patients who are considered to be inappropriate to the subject of this study by the investigator.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2008-09; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Takizawa, MD, Study Chair — Cancer Institute Hospital; Toshiharu Kamura, MD, Study Chair — Yanagawa Hospital; Ting-Chang Chang, MD, Study Chair — Chang Gung Memorial Hospital; Soon-Beom Kang, MD, Study Chair — Konkuk University Medical Center
Locations (4):
- Japan (2):
  - Yanagawa Hospital, Chikushimachi, Yanagawa, Fukuoka
  - Cancer Institute Hospital, Ariake, Koto-ku, Tokyo
- Konkuk University Medical Center, Hwayang-dong, Gwangjin-gu, Seoul, South Korea
- Chang Gung Medical Foundation- Linkou, Fu-Hsing Saint Kuei Shan Hsiang, TaoYuan Hsien, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 375 patients were randomized to Arm A (189) or Arm B (186); of these, 364 patients(188 and 176, respectively) received study treatment. 11 patients (1 and 10, respectively) did not receive allocated intervention because of 'withdrew consent(1 and 6, respectively)' , 'ineligible criteria(3 in Arm B)', or 'investigator's discretion(1 in Arm B)'.
Period: Overall Study
Arm/Group | S-1 + Cisplatin (Arm A) | Cisplatin (Arm B)
Started | 188 | 176
Completed | 188 | 176
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 364 (188 in Arm A; 176 in Arm B) received study treatment. Two patients in Arm B were excluded in the efficacy analysis, because of insufficient informed consent, and missing efficacy data.
Groups:
- Total: Total of all reporting groups
Arm/Group | S-1 + Cisplatin (Arm A) | Cisplatin (Arm B) | Total
Number analyzed (Participants) | 188 | 174 | 362
Age, Continuous [Median (Full Range); unit: years] | 55 [27 to 84] | 52.5 [28 to 81] | 54 [27 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 174 | 362
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 52 | 49 | 101
  Japan | 110 | 105 | 215
  Taiwan | 26 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: From the date of randomization to death from any cause, assessed up to 296 events or the end of November 2015, whichever was earlier, each three months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1 + Cisplatin (Arm A) | Cisplatin (Arm B)
Number analyzed (Participants) | 188 | 174
months | 21.9 [18.6 to 25.8] | 19.5 [17.0 to 24.3]
Statistical Analysis 1: Comparison: S-1 + Cisplatin (Arm A); Test type: Superiority; p = 0.125, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.05]

2. Secondary Outcome: Progression Free Survival, Safety
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: About Progression free survival, from the randomization to disease progression or death, whichever came first, assessed up to until primary outcome came each three months, and about safety, from the first treatment to 30 days after the last treatment
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1 + Cisplatin (Arm A) | Cisplatin (Arm B)
Number analyzed (Participants) | 188 | 174
months | 7.3 [6.7 to 8.1] | 4.9 [4.4 to 5.7]
Statistical Analysis 1: Comparison: S-1 + Cisplatin (Arm A); Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.48 to 0.80]

ADVERSE EVENTS:
Time Frame: From the date of the first treatment to 30 days after the last treatment
Description: A total of 364 (188 in Arm A; 176 in Arm B) received study treatment. One patient in Arm B were excluded in the safety analysis, because of insufficient informed consent.
Arm/Group | S-1 + Cisplatin (Arm A) | Cisplatin (Arm B)
All-Cause Mortality (participants affected / at risk) | 7/188 | 3/175
Serious Adverse Events (participants affected / at risk) | 72/188 | 34/175
Other Adverse Events (participants affected / at risk) | 188/188 | 172/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S-1 + Cisplatin (Arm A) (N=188) | Cisplatin (Arm B) (N=175)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascities (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Illeus (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 0
Disease progression (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Infective myositis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 5 | 4
Ureteritis (Infections and infestations) | 0 | 1
Uterine infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Blood uric acid decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 10 | 5
Neutrophil count decreased (Investigations) | 12 | 0
Platelet count decreased (Investigations) | 5 | 0
White blood cell count decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Hydroneprosis (Renal and urinary disorders) | 2 | 2
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 2
Ureteric obstruction (Renal and urinary disorders) | 5 | 2
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Breast engorgement (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombosis (Vascular disorders) | 10 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S-1 + Cisplatin (Arm A) (N=188) | Cisplatin (Arm B) (N=175)
Abdominal distension (Gastrointestinal disorders) | 12 | 5
Abdominal pain (Gastrointestinal disorders) | 29 | 26
Abdominal pain upper (Gastrointestinal disorders) | 24 | 9
Constipation (Gastrointestinal disorders) | 61 | 48
Diarrhoea (Gastrointestinal disorders) | 94 | 51
Dyspesia (Gastrointestinal disorders) | 21 | 12
Gastritis (Gastrointestinal disorders) | 19 | 10
Nausea (Gastrointestinal disorders) | 153 | 134
Stomatitis (Gastrointestinal disorders) | 59 | 16
Vomiting (Gastrointestinal disorders) | 103 | 71
Fatigue (Gastrointestinal disorders) | 109 | 79
Influenza like illness (General disorders) | 29 | 17
Oedema peripheral (General disorders) | 41 | 16
Pyrexia (General disorders) | 38 | 20
Localised oedema (General disorders) | 20 | 15
Hypersensitivity (Immune system disorders) | 10 | 9
Cystitis (Infections and infestations) | 12 | 9
Upper respiratory tract infection (Infections and infestations) | 12 | 6
Urinary tract infection (Infections and infestations) | 17 | 12
Alanine aminotransferase increased (Investigations) | 38 | 23
Aspartate aminotransferase increased (Investigations) | 33 | 15
Blood albumin decreased (Investigations) | 46 | 23
Blood bilirubin decreased (Investigations) | 21 | 3
Blood calcium decreased (Investigations) | 18 | 6
Blood creatinine increased (Investigations) | 38 | 39
Blood potassium decreased (Investigations) | 39 | 9
Blood sodium decreased (Investigations) | 30 | 15
Haemoglobin decreased (Investigations) | 147 | 87
Lymphocyte count decreased (Investigations) | 21 | 10
Neutrophil count decreased (Investigations) | 148 | 65
Platelet count decreased (Investigations) | 90 | 26
Weight decreased (Investigations) | 38 | 10
Weight increased (Investigations) | 11 | 10
White blood cell count decreased (Investigations) | 92 | 52
Protein urine present (Investigations) | 29 | 13
Decreased appetite (Metabolism and nutrition disorders) | 141 | 105
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 10
Dizziness (Nervous system disorders) | 37 | 15
Dysgeusia (Nervous system disorders) | 34 | 12
Headache (Nervous system disorders) | 32 | 31
Peripheral sensory neuropathy (Nervous system disorders) | 39 | 22
Insomnia (Psychiatric disorders) | 28 | 21
Ureteric obstruction (Renal and urinary disorders) | 10 | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 11 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 48 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 36 | 18
Thrombosis (Vascular disorders) | 14 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other